CLINICAL TRIAL: NCT06747832
Title: A Single-center, Single-arm Clinical Study of the Efficacy and Safety of INK Cells As Maintenance Therapy After Chemoradiotherapy for Small Cell Lung Cancer
Brief Title: INK Cells As Maintenance Therapy After Chemoradiotherapy for Small Cell Lung Cancer
Acronym: iNK-SCLC
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangzhou Ruixin Biotechnological Co., LTD (Industry)
Collaborators: Weifang People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iNK-SCLC
Record Dates: First submitted 2024-12-08; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Small Cell Lung Cancer
Keywords: iNK Cellular therapy sclc
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: A single-center, single-arm clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- iNK Cell therapy group (Experimental): Intravenous infusion of iNK cells is given to the subject, 5*108 to 1*109 cells/dose, three doses per week, a total of 6 doses. And then 1*109 cells/dose, one doses every 4 weeks , a total of 5 doses.
  Interventions: Drug: iNK cells

INTERVENTIONS:
Drug: iNK cells — Intravenous infusion of iNK cells is given to the subject, 5*108 to 1*109 cells/dose, three doses per week, a total of 6 doses. And then 1*109 cells/dose, one doses every 4 weeks , a total of 5 doses.

SUMMARY:
This is a clinical study on the use of iNK cells for the treatment of small cell lung cancer.

DETAILED DESCRIPTION:
Natural killer (NK) cells are lymphocytes of the innate immune system and could recognize and kill a wide range of cells in distress, particularly tumour cells and cells infected with viruses. Induced pluripotent setm cells(iPSCs) derived NK cells have better proliferative capacity and homogeneity than donor peripheral blood or umbilical cord blood derived NK cells. The investigators conduct this clinical study to evaluate the efficacy and safety of INK cells as maintenance therapy after chemoradiotherapy for small cell lung cancer and The purpose of investigators is to find new treatment option.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
2. Age ≥18 years old and ≤ 75 years old at the time of signing the ICF
3. Have cytologically or histologically confirmed diagnosis for the patients with locally advanced unresectable or metastatic small cell lung cancer.
4. Have measurable disease as assessed by the investigator according to RECIST 1.1.
5. Have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
6. Have a life expectancy of ≥ 3 months.
7. Female participants: Women of childbearing potential (WOCBP) must use a highly effective form of contraception from the screening visit until at least 12 months after the final dose of iNK cells.
8. Male participants: Males must be sterile (biologically or surgically) or use a highly effective method of contraception from the screening visit until at least12 months after the final dose of iNK cells.

Exclusion Criteria:

1. Has evidence of insufficient organ function. 1.1 Has active or clinically significant cardiac disease including: 1.1.1 Severe heart rhythm or conduction abnormalities, corrected QT interval (QTc) ≥ 480 ms.

   1.1.2 Complete left bundle branch block, second- or third-degree atrioventricular block.

   1.1.3 Severe, uncontrolled cardiac arrhythmias requiring medication. 1.1.4 New York Heart Association (NYHA) class II or above congestive heart failure.

   1.1.5 Left ventricular ejection fraction (LVEF) < 50% in color Doppler echocardiography.

   1.1.6 History of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, severe pericardial disease, ECG evidence of acute ischemic or active conduction system abnormalities within 6 months prior to recruitment.

   1.2 Renal: SCR > 1.5 x ULN or calculated creatinine clearance (Cockcroft-Gault Formula) <60 mL/min.

   1.3 Liver: 1.3.1 total bilirubin > 1.5 x ULN. 1.3.2 AST>2x ULN or ALT>2x ULN. AST/ALT can be as high as 5× ULN in liver metastases, but it cannot be accompanied by elevated bilirubin 1.4 lung:

   > grade 1 dyspnea and oxygen saturation ≤ 91% in non oxygen breathing state. 1.5 Hematological: 1.5.1 Absolute neutrophil count (ANC) < 1.5 x 109/L. 1.5.2 Platelet count< 100 x 109/L. 1.5.3 Hemoglobin < 9.0g/dL. 1.5.4 International normalized ratio (INR) > 1.5 times ULN, and activated partial prothrombin time (APTT) > 1.5 times ULN;
2. At the time of screening, patients with symptomatic central nervous system (CNS) metastases (asymptomatic CNS metastases, or asymptomatic after local treatment and stable condition for 4 weeks can be enrolled).
3. Those with a history of central nervous system before screening, such as epilepsy, cerebral ischemia / hemorrhage, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, cerebral organic syndrome, mental disease or any autoimmune disease involving the central nervous system.
4. Those who stopped systemic hormone therapy for less than 72 hours before cell transfusion; But it is allowed to use a physiological substitute amount of hormone (such as prednisone < 10mg / D or equivalent).
5. Active systemic autoimmune disease is known before screening and is under treatment.
6. 8. Those who meet any of the following conditions during screening: 6.8.1 Positive for hepatitis B surface antigen (HBsAg) and / or hepatitis B e antigen (HBeAg).

   6.8.2 Hepatitis B e antibody (HBE AB) and / or hepatitis B core antibody (HBC AB) are positive, and the copy number of HBV-DNA is greater than the lower measurable limit.

   6.8.3 Positive for hepatitis C antibody (HCV AB). 6.8.4 Positive anti Treponema pallidum antibody (TP AB). 6.8.5 HIV antibody test positive. 6.8.6 The copy number of EBV-DNA and cmv-dna is greater than the lower measurable limit.
7. Participated in other intervention clinical studies within 4 weeks before screening;
8. People who are allergic to human blood albumin.
9. People who are allergic to IL-2.
10. Patients who are judged by the investigator to be unsuitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Event (AE) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v5.0 | 12 months
Objective-response rate (ORR) | 12 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 12 months
Duration of Response (DoR) | 12 months
Overall Survival (OS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yu Guohua Guohua Yu, Director of the Cancer Dpartment, Study Chair — Weifang People's Hospital
Locations (1):
- Weifang People's Hospital, Weifang, Shandong Province, China., China

IPD SHARING:
Plan to Share IPD: Yes
What data in particular will be shared? Individual participant data that underlie the results reported in this article, after deidenti- fication (text, tables, figures, and appendices).
  What other documents will be available？ Study Protocol. When will data be available (start and end dates)? Beginning 9 months and ending 36 months following article publication. With whom? Investigators whose proposed use of the data has been approved by an independent review committee(learned intermediary) identified for this purpose.
  For what types of analyses? For individual participant data meta-analysis. By what mechanism will data be made available? Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in clinical research center of the fifth affiliated hospital of Guangzhou medical university (https://www.wfph.cn/news/44/).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee(learned intermediary) identified for this purpose.